CLINICAL TRIAL: NCT01955356
Title: Evaluation of Induced Endometrial Injury in the Subsequent IVF Cycle.
Brief Title: Embryo Implantation After Induced Endometrial Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Collaborators: IVI Madrid (Other); IVI Barcelona (Other); IVI Murcia (Other); Vida Recoletas Sevilla (Other); IVI Bilbao (Other); IVI Vigo (Other); Instituto Valenciano de Infertilidad, IVI Alicante (Other)
Responsible Party: Principal Investigator, Carmina Vidal, MD, Obstetrics and Gynecology, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1306-C-119-CV/IVI Valencia
Record Dates: First submitted 2013-09-28; First posted 2013-10-07 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Sterility
Keywords: Scratching; Endometrial biopsy; Ongoing embryo implantation; Assisted reproductive techniques
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scratching (Experimental): induced endometrial injury
  Interventions: Procedure: Scratching
- No scratching (No Intervention): None intervention

INTERVENTIONS:
Procedure: Scratching — Endometrial biopsy
  Other Names: Endometrial induced injury
  Arms: Scratching

SUMMARY:
Some studies have revealed that an induced endometrial injury could improve embryo human implantation in patients with implantation failure.

The purpose of this study is to determine whether the induced endometrial injury could be beneficial for regular patients undergoing IVF

DETAILED DESCRIPTION:
Endometrial induced injury has been suggested that could improve embryo implantation in cases of patients with recurrent implantation failure. The mechanisms that induce that improvement remain unknown.

We want to analyse if the endometrial induce injury could be useful in cases of standard patients who require assisted reproductive techniques.

For that purpose we will start a randomized controlled trial with the ideal background in implantation in ART, the egg donation programme.

ELIGIBILITY:
Inclusion Criteria:

* 19-44 aged women
* 19-29.9 Kg/m2.
* 1st or 2nd fresh embryo transfer ( egg donation).
* 1 or 2 blastocysts available.
* written agreement.
* > or = 6 mms endometrial thickness.

Exclusion Criteria:

* Premature ovarian failure.
* Endometrial pathology.
* Insufficient endometrial development.
* Hydrosalpinx
* Mullerian malformations.

Ages: 19 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Ongoing implantation rate (OIR) | 12 weeks of pregnancy

SECONDARY OUTCOMES:
Live born rate (LBR) | 9 months after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Carmina Vidal, MD, Principal Investigator — IV VALENCIA
Locations (1):
- IVI Valencia, Valencia, Spain